CLINICAL TRIAL: NCT00899574
Title: Phase II Evaluation of Imiquimod, a Topical Toll-like Receptor 7 (TLR7) Agonist in Breast Cancer Patients With Chest Wall Recurrence or Skin Metastases
Brief Title: Imiquimod for Breast Cancer Patients With Chest Wall Recurrence or Skin Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU 09-0225
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: toll-like receptor; toll-like receptor agonist; recurrent breast cancer; breast cancer metastasized to skin and/or chestwall; immunomodulator
MeSH Terms: conditions — Breast Neoplasms | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imiquimod (Experimental): Each treatment cycle consists of 8 weeks.
  Weeks 1-8: day 1-5 of each week: 1 packet imiquimod 5% cream applied overnight, day 6-7 of each week: rest period.
  Patients with responding or stable local disease (non-progressors) may continue to receive treatment following the same schedule (as outlined above for the first cycle) until complete tumor regression, unacceptable toxicity or progression of disease.
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Imiquimod — Each treatment cycle consists of 8 weeks.
  Weeks 1-8: day 1-5 of each week: 1 packet imiquimod 5% cream applied overnight, day 6-7 of each week: rest period.
  Patients with responding or stable local disease (non-progressors) may continue to receive treatment following the same schedule (as outlined above for the first cycle) until complete tumor regression, unacceptable toxicity or progression of disease.
  Other Names: Aldara

SUMMARY:
The purpose of this trial is to determine the safety and efficacy of Imiquimod, a Toll-like receptor 7 agonist in breast cancer (for chestwall recurrences or metastases to the skin).

DETAILED DESCRIPTION:
TLR agonists are novel agents for cancer therapy which modify the immune response. Imiquimod, a synthetic TLR7 agonist has proven immunomodulatory activity when applied topically, leading to clearance of human papilloma virus (HPV)-induced genital warts and primary skin malignancies. Its effects will now be examined in breast cancer metastatic to the skin. If effective, it will add a relatively non-toxic approach to the treatment armamentarium for this patient population frequently resistant to conventional therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-confirmed breast cancer (prior histological documentation is acceptable).
* Patients with measurable skin metastases (chest wall recurrence and/or non-chest wall skin metastases are eligible).
* Skin metastases not suitable for or patient refusing definitive surgical resection and radiation.
* (Cohort 1) Concurrent systemic cancer therapy (hormones, biologics or chemotherapy) is allowed if distant metastases have been non-progressing (stable or responding) on that regimen for > or = 12 weeks and skin metastases are non-responsive (stable or progressing) as assessed by the investigator.

(Cohort 2) Any concurrent systemic therapy is allowed

* Age at least 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status < or = 2.
* Patients must have biopsy-accessible tumor (skin metastases) and agree to biopsies required by protocol.
* Patients must have adequate organ and bone marrow function as defined below:

  * absolute neutrophil count > or = 1,500/microliter
  * hemoglobin > or = 9.5 grams/deciliter
  * platelets >or = 75,000/microliter
  * total bilirubin < or = 1.5 X institutional upper limit of normal
  * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) < or = 2.5X institutional upper limit of normal
  * creatinine < or = 1.5 X institutional upper limit of normal
* Informed consent.

Exclusion Criteria:

* Brain metastases unless resected or irradiated and stable > or = 8 weeks.
* Treatment with other investigational agents.
* Patients who have received radiotherapy, high-potency corticosteroids, intralesional therapy, laser therapy or surgery other than biopsy to the target area within 4 weeks prior to first dosing of study agent.
* Patients who have received hyperthermia to the target area within 10 weeks prior to first dosing of study agent.
* Patients with an uncontrolled bleeding disorder.
* Patients who will be therapeutically anticoagulated with heparins or coumadin at the time of the biopsy (they are eligible if anticoagulation can be held prior to biopsy as per investigator). Patients on aspirin and other platelet agents are eligible.
* Patients with known immunodeficiency or receiving immunosuppressive therapies.
* History of allergic reactions to imiquimod or its excipients.
* Uncontrolled intercurrent medical illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy or lactation.
* Women of childbearing potential not using a medically acceptable means of contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Adams, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Institute, New York, New York, United States

REFERENCES:
- [Result] Adams S, Kozhaya L, Martiniuk F, Meng TC, Chiriboga L, Liebes L, Hochman T, Shuman N, Axelrod D, Speyer J, Novik Y, Tiersten A, Goldberg JD, Formenti SC, Bhardwaj N, Unutmaz D, Demaria S. Topical TLR7 agonist imiquimod can induce immune-mediated rejection of skin metastases in patients with breast cancer. Clin Cancer Res. 2012 Dec 15;18(24):6748-57. doi: 10.1158/1078-0432.CCR-12-1149. Epub 2012 Jul 5. PMID 22767669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten patients were enrolled to this study between Nov. 2009 and Nov. 2010 at New York University Medical Center and affiliated hospital.
Period: Overall Study
Arm/Group | Imiquimod
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imiquimod
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 50 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Clinical Response+ Partial Response)
Description: This is defined as percentage of patients who achieved complete clinical response or partial response at end of cycle 1 of treatment. The tumor size will be measured as lesion surface area (region of interest, ROI). The response to the treatment is then evaluated as a function of post-treatment over pre-treatment ROI, expressed in percentage. Response criteria for this study are based on European Organisation for Research and Treatment of Cancer definitions for chest wall tumors: complete clinical response: absence of any detectable residual disease; partial response: <50% of ROI change.
Time Frame: 9 weeks
Population: Patients who completed 1 cycle of treatment (8 weeks) and response evaluation at week 9.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Imiquimod
Number analyzed (Participants) | 10
percentage of patients | 20 [3 to 56]

2. Secondary Outcome: Clinical Benefits
Description: This outcome measure is defined as number of patients with improvement of symptoms after 8 weeks of treatment.
Time Frame: 9 weeks
Population: Patients who completed 1 cycle of treatment (8 weeks) and response evaluation at week 9.
Measure: Number; unit: patients
Arm/Group | Imiquimod
Number analyzed (Participants) | 10
patients
  Pain improvement | 4
  Pruritus improvement | 5
  Dermatology Life Quality Index (DLQI) improvement | 0

ADVERSE EVENTS:
Time Frame: Up to 18 weeks.
Arm/Group | Imiquimod
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod (N=10)
Anorexia (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Distension/Bloating, Abdominal (Gastrointestinal disorders) | 1 (2)
Edema: Limb (Blood and lymphatic system disorders) | 1 (1)
Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 1 (1)
Fever (In The Absence Of Neutropenia, Where Neutropenia Is Defined As Anc <1.0 X 10e9/L) (General disorders) | 1 (1)
Flu-Like Syndrome (General disorders) | 1 (1)
Hemorrhage/Bleeding - Other (General disorders) | 1 (1)
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils (Infections and infestations) | 1 (1)
Mood Alteration (Nervous system disorders) | 1 (6)
Nausea (Gastrointestinal disorders) | 2 (8)
Neurology - Other (Nervous system disorders) | 1 (1)
Neuropathy: Sensory (Nervous system disorders) | 1 (8)
Pain (General disorders) | 6 (33)
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 3 (6)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 3 (6)
Rash: Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1 (2)
Rigors/Chills (General disorders) | 2 (2)
Skin Breakdown/Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Weight Loss (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The 20% response rate would have justified to continue; but the study was concluded and a new trial of imiquimod and local radiotherapy (NCT01421017) is open, based on preclinical findings indicating that the combination was more effective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes